CLINICAL TRIAL: NCT00922818
Title: Clinical Outcomes for Anatomic Nerve Sparing Radical Perineal Prostatectomy
Brief Title: Study of Anatomic Nerve Sparing Radical Perineal Prostatectomy
Acronym: RPP
Status: Withdrawn | Type: Observational
Why Stopped: recruitment issues
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-05-VA02
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2018-08-20 (Actual); Status verified 2018-08

CONDITIONS: Prostate Cancer
Keywords: Perineal; Prostatectomy; Nerve; Anatomic; Surgery; Neoplasms, Prostatic; Prostate Cancer; Prostate Neoplasms; Prostatic Cancer; Prostate; Cancer; Recurrent
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Radical perineal prostatectomy patients: Radical perineal prostatectomy patients

SUMMARY:
Our objective is to evaluate the clinical outcomes for the anatomic radical perineal prostatectomy (RPP) for the surgical management of prostate cancer. We will report the perioperative, oncologic, and functional outcomes in patients undergoing the radical perineal prostatectomy at our institution.

DETAILED DESCRIPTION:
The purpose of our study is to evaluate perioperative, oncologic, and functional outcomes for the anatomic radical perineal prostatectomy. The anatomic radical perineal prostatectomy is standard-of-care surgical approach to the surgical management of localized prostate cancer. The operative technique selected for radical prostatectomy is largely based on patient preference after appropriate counseling, and surgeon recommendation based on surgical considerations and surgeon experience. Outcome data for the anatomic radical perineal prostatectomy will represent a valuable addition to the published body of literature. Our study is a prospective clinical outcome data collection and analysis and we will be looking at data within several domains. First, perioperative data will be collected to evaluate the OR time, blood loss, surgical complications, and length of hospital stay for the anatomic radical perineal prostatectomy. Second, oncologic efficacy of this procedure will be reported, based on margin status of surgical specimens, which will be correlated with tumor features (Gleason score, tumor volume, pre-op PSA score). Third, functional outcomes will be evaluated by comparing urinary, sexual, and bowel function in the pre-op and post-op settings. This third domain will be accomplished by employing the following validated questionnaires (attached - SHIM, IPSS, and EPIC-26). These questionnaires will be filled out at 3 time-points: pre-op, and at 3 months and 12 months post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Perineal prostatectomy for prostate cancer at Maimonides Medical Center

Exclusion Criteria:

* Dementia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing anatomic perineal prostatectomy at Maimonides Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05-26 (Actual); Study Completion 2011-05-26 (Actual)

PRIMARY OUTCOMES:
Surgical margin-free rate | June 2011
  proportion of negative margins

SECONDARY OUTCOMES:
EPIC-26 Functional Outcome Status | June 2011
  validated outcome questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jason B. Wynberg, MD, FACS, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

REFERENCES:
- See also: Prostate Cancer Information — http://www.nlm.nih.gov/medlineplus/prostatecancer.html
- See also: Perineal Anatomy — http://en.wikipedia.org/wiki/Perineum